CLINICAL TRIAL: NCT05899790
Title: The Effect of Information About the Operating Room Environment With Virtual Reality Glasses on the Anxiety Level and Vital Findings of the Patients: A Randomized Controlled Study
Brief Title: The Effect of Information About the Operating Room Environment With Virtual Reality Glasses on the Anxiety Level
Acronym: VRanxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Serpil ÇağlIyan payas, lecturer, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Eastern MU-SBF-HB-SÇP-01
Record Dates: First submitted 2022-03-30; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Preoperative Anxiety
Keywords: Preoperative anxiety,; virtual reality,; abdominal surgery,; information about the operating room environment

STUDY DESIGN:
Intervention Model Description: 2 Group
  1. İntervention
  2. Control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Forty patients who received standard care in the pre-abdominal surgery clinic and preoperative waiting area will form the control group.
- intervention group (Experimental): In addition to standard care, 40 patients who were informed about the SG application and the operating room environment will form the intervention group.
  Interventions: Other: VR

INTERVENTIONS:
Other: VR — The first interview with the patients in the intervention group will be held in the afternoon, the day before the surgery. After completing the forms and scale the video containing information about the operating room environment will be applied to the patients through SG glasses and headphones.
  Before the surgical intervention, patients admitted to the pre-operative waiting area from the clinic, the video containing information about the operating room environment will be watched by the patients through SG glasses and headphones.
  Other Names: Virtual reality
  Arms: intervention group

SUMMARY:
Virtual Reality (VR) applications, one of the commonly emphasized approaches in the medical field recently, is in place as an intervention method applicable in various fileds of medicine for distraction, experiencing being exposed to events creating stress and palliating anxiety through providing materials which may distract the patient's attention from a stressful condition. The study has been planned in order to evaluate the effect of the notification regarding the theatre environment through virtual reality to the patients, who are to go through abdominal surgical intervention, on the anxiety level and the vital signs during the surgical intervention.

Being a non-pharmacological clinical randomize controlled one, the study shall be conducted in Dr. Burhan Nalbantoğlu State Hospital of TRNC Ministry of Health surgical service and preoperative waiting area.

Sample number has been determined through power analysis using G*Power 3.1.9.2 software. Taking (2017) "The effect of virtual reality in reducing preoperative anxiety in patients prior to arthroscopic knee surgery: A randomised controlled trial" study of Robertson and friends as the reference, the effect size, regarding the anxiety scores of experiment and control groups participants, has been determined as 0,63. Accordingly, sample size has been calculated as 71 people necessary for 95% (1-β=0,95) power at d=0,63 and α=0,05 levels. Taking into account there may be losses during the study, it has been planned to involve 80 people, so as to have 40 people per each group, in the study.

Since the patients, who are to be involved in the study, are not known; in order to assign same quantity of patients to each group prior to the study, randomization shall be done through using block randomization technique in GraphPad software so as to have 40 patients in the intervention group and 40 in the control group. The patients who receive standard clinical care prior to abdominal surgical intervention shall constitute the control group, the patients who receive information about operating room environment through VR goggles in addition to standard clinical care shall constitute the intervention group. The data shall be collected through "Individual characteristics Form", ''Patient Charts'', ''Surgical Anxiety Scale'', ''Galvanic Skin Sensor (GSS) Measurement Table''.

SPSS 26 Statistical analysis program shall be used for evaluating the study data. The acquired data shall be tested at 95% confidence interval, p<0,05 level of significance. Number, percentage distributon and standard deviation for the definitive data analysis, chi square test for experiment and control groups' basic particulars similarity, Shapiro-Wilk for normality analysis of dependent variables, Student t test or Annova for the comparison of pre-test and final test scores of experiment control groups, the comparisons of variables giving normal distribution among the groups as per the normal distributon in the comparison of experiment control groups' pre-test and final test scores, Mann Whitney U test or Kruskal Wallis test for the variables of non-normal distribution shall be used.

DETAILED DESCRIPTION:
Surgical interventions, which are widely used for health improvement and disease treatment, are one of the most important experiences in an individual's life. Surgical interventions, regardless of simple or life threatening, turn in to a condition leading to individual's loss of control on his body for a limited time and anxiety due to not having sufficient information about the subject although they are positive things which would provide recovery from illness. It is known that more medical complications build up in patients who have higher level of anxiety during the medical process. Although the factors, which trigger the anxiety, vary significantly among the individuals, the effects of common or lasting anxiety cases are usually similar. These factors may lead to effects such as pain, sinus tachycardia, hypertension, cardiac arrhythmia, surgical interventions, increase in anesthesia and analgesia necessities, latency in wound healing and discharge periods. Operating rooms being complex and unusual environments and getting anesthesia lead to anxiety and fear in patients. Since focusing on pharmacological intervetions in the current management of anxiety increases complications, which may build up inthe patient; easy to use, noninvasive non-pharmacological applications are required. Virtual Reality (VR) applications, one of the commonly emphasized approaches in the medical field recently, is in place as an intervention method applicable in various fileds of medicine for distraction, experiencing being exposed to events creating stress and palliating anxiety through providing materials which may distract the patient's attention from a stressful condition. The study has been planned in order to evaluate the effect of the notification regarding the theatre environment through virtual reality to the patients, who are to go through abdominal surgical intervention, on the anxiety level and the vital signs during the surgical intervention.

Being a non-pharmacological clinical randomize controlled one, the study shall be conducted in Dr. Burhan Nalbantoğlu State Hospital of TRNC Ministry of Health surgical service and preoperative waiting area. The criteria for being involved in the study have been defined as patients who are of 18 years old and over, are to go through abdominal surgical intervention, are conscious, have orientation of place-person and time, do not have any visual, audial or mental problem, have the ability of understanding the instructions of the study and reacting, can communicate in Turkish and give written approval for participating in the study. The criteria of being excluded form the study have been defined as the patients who regularly receive phytotherapy or pharmacotherapy for anxiety, are diagnosed with hypertension, cardiac arrhythmia, have facial injuries preventing comfortable utilization of VR hardware and are unpremedicated. The criteria of elimination from the study shall be composed of the patients who want to quit at own request, can not comply with the study process and conditions.

Sample number has been determined through power analysis using G*Power 3.1.9.2 software. Taking (2017) "The effect of virtual reality in reducing preoperative anxiety in patients prior to arthroscopic knee surgery: A randomised controlled trial" study of Robertson and friends as the reference, the effect size, regarding the anxiety scores of experiment and control groups participants, has been determined as 0,63. Accordingly, sample size has been calculated as 71 people necessary for 95% (1-β=0,95) power at d=0,63 and α=0,05 levels. Taking into account there may be losses during the study, it has been planned to involve 80 people, so as to have 40 people per each group, in the study.

Since the patients, who are to be involved in the study, are not known; in order to assign same quantity of patients to each group prior to the study, randomization shall be done through using block randomization technique in GraphPad software so as to have 40 patients in the intervention group and 40 in the control group. The patients who receive standard clinical care prior to abdominal surgical intervention shall constitute the control group, the patients who receive information about operating room environment through VR goggles in addition to standard clinical care shall constitute the intervention group. The data shall be collected through "Individual characteristics Form", ''Patient Charts'', ''Surgical Anxiety Scale'', ''Galvanic Skin Sensor (GSS) Measurement Table''.

SPSS 26 Statistical analysis program shall be used for evaluating the study data. The acquired data shall be tested at 95% confidence interval, p<0,05 level of significance. Number, percentage distributon and standard deviation for the definitive data analysis, chi square test for experiment and control groups' basic particulars similarity, Shapiro-Wilk for normality analysis of dependent variables, Student t test or Annova for the comparison of pre-test and final test scores of experiment control groups, the comparisons of variables giving normal distribution among the groups as per the normal distributon in the comparison of experiment control groups' pre-test and final test scores, Mann Whitney U test or Kruskal Wallis test for the variables of non-normal distribution shall be used.

ELIGIBILITY:
Inclusion Criteria:

* who are of 18 years old and over,
* are to go through abdominal surgical intervention,
* are conscious, have orientation of place-person and time,
* do not have any visual,
* audial or mental problem,
* have the ability of understanding the instructions of the study and reacting,
* can communicate in Turkish
* and give written approval for participating in the study

Exclusion Criteria:

* the patients who regularly receive phytotherapy or pharmacotherapy for anxiety,
* are diagnosed with hypertension,
* cardiac arrhythmia,
* have facial injuries preventing comfortable utilization of VR hardware
* and are unpremedicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Surgical Anxiety Scale | two day
  maximum: 4 minimum: 0

CONTACTS AND LOCATIONS:
Overall Officials: serpil çağlıyan payas, lecturer, Principal Investigator — DOĞU AKDENİZ ÜNİVERSİTESİ
Locations (1):
- Doğu Akdeniz Üniversitesi, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/33036555/
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/32247709/
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/34252034/